CLINICAL TRIAL: NCT00582647
Title: Collection of Tissue, Blood and Other Specimens From Patients With Benign and Malignant Tumors of the Soft Tissue, Gastrointestinal Tract, and Other Intra-abdominal Sites.
Brief Title: Collection of Tissue & Blood From Patients w/ Benign & Malignant Tumors of the Soft Tissue & Gastrointestinal Tract
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-032
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer; Bile Duct Neoplasms; Gastric Cancer; Liver Cancer; Melanoma; Pancreatic Cancer; Sarcoma
MeSH Terms: conditions — Esophageal Neoplasms; Bile Duct Neoplasms; Stomach Neoplasms; Liver Neoplasms; Melanoma; Pancreatic Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, Blood, Peritoneal, Pleural, Cyst, and Other gastrointestinal fluid

SUMMARY:
Doctors at Memorial Sloan Kettering Cancer Center and at other institutions study normal and cancer cells. To study these cells we need to have human tissue, body fluids, and blood. The patient will be having or have had a procedure to remove tissue. The doctors would like to use some of this tissue. The doctors will use it for laboratory studies on the causes, prevention, diagnosis and treatment of sarcoma, gastrointestinal or other intra-abdominal cancers. They will only use extra tissue left over after all needed testing has been done. They would also like to study components of the immune blood cells and blood serum (the liquid portion of the blood). In some patients they will take a blood sample before the tissue or body fluid is removed, usually at the same time that other routine pre-procedure blood tests are drawn. If thet need more blood, it will be drawn when the patient is seeing the doctor anyway. We will not draw more than 50cc (4-5 tablespoons) at any one time. With the patient's permission, thet may also send a small portion of the blood and/or a sample of the tissue to a repository at the National Cancer Institute. This will be used to identify special proteins in the blood or tissue that may be useful for diagnosing cancer. Information about the treatment and the response to treatment may be linked to the tissue specimens obtained. This information may be important for the research studies that will be done on the tissue, body fluid and blood specimens. All of this information will be kept in strictest confidence; they will use it only for biomedical research. The patient's name will not be used in any report.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* All patients with benign or malignant tumors of the soft tissues, gastrointestinal tract, and other intra-abdominal sites who will have or have had tissue, peritoneal, pleural, cyst, urine, and/or other gastrointestinal fluid removed for therapeutic or diagnostic purposes.
* Patients will be entered without preference for any particular racial/ethnic group.
* Patients may have received prior hormonal therapy, cytotoxic chemotherapy, irradiation, immunotherapy or surgical therapy.
* Tissue and body fluid specimens must be a large enough quantity to allow routine pathological analysis, with the research laboratory specimen removed from the residual specimen which would otherwise be discarded.

Healthy Control Subjects:

* Any male or female with no concurrent malignancies (except for localized basal cell or squamous cell skin cancer) within 5 years of enrollment.
* > or = to 18 years of age
* Any MSKCC employee will be allowed to participate as a healthy control, provided they fulfill the above inclusion criteria and they enroll willfully and voluntarily

Exclusion Criteria:

Healthy Control Subjects:

* Attending physicians authorized to obtain informed consent may exercise discretion in excluding individuals for appropriate medical or other (e.g. mentally impaired) reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2000-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To obtain & store tissues, blood, peritoneal, pleural, cyst & other gastrointestinal fluid from patients with benign or malignant tumors in order to carry out future laboratory studies on the causes, prevention, diagnosis & treatment of certain cancers. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kingham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org